CLINICAL TRIAL: NCT03453866
Title: Effect of Warmed Irrigation Fluid on Immediate Post-operative Pain Scores in Patients Undergoing Hip Arthroscopy
Brief Title: Effect of Warmed Irrigation in Hip Arthroscopy Undergoing Hip Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-2399
Record Dates: First submitted 2018-02-14; First posted 2018-03-05 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Femoro Acetabular Impingement; Pain, Postoperative
Keywords: Hip Arthroscopy; Warmed Fluids
MeSH Terms: conditions — Femoracetabular Impingement; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Controlled Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Sealed Opaque Envelope
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warmed Arthroscopic Fluids (Experimental): Arthroscopic Fluids will be warmed to 38 degrees Celsius during procedure with active warming device. Temperature will be measured in real time.
  Interventions: Procedure: Warmed Arthroscopic Fluids
- Room Temperature Arthroscopic Fluids (Active Comparator): Arthroscopic fluids will be kept at room temperature and will not be warmed per current standard of care. Temperature will be measured in real time.
  Interventions: Procedure: Room Temperature Arthroscopic Fluids

INTERVENTIONS:
Procedure: Warmed Arthroscopic Fluids — Warmed Arthroscopic Fluids
  Arms: Warmed Arthroscopic Fluids
Procedure: Room Temperature Arthroscopic Fluids — Room Temperature Arthroscopic Fluids
  Arms: Room Temperature Arthroscopic Fluids

SUMMARY:
The purpose of this study is to determine if pre-warming of arthroscopic fluid reduces immediate post-surgical pain in hip arthroscopy patients. The investigators hypothesize there will be a significant decrease in the Visual Analog Score (VAS) measured 30 minutes post-operatively in the warmed fluid group compared to the control group. Secondary outcome measures to be collected will include VAS scores 60 minutes after surgery and on post-operative day (POD) one. Additionally, the investigators will collect post-operative temperature measured 30 and 60 minutes post-operatively as well as morphine equivalent dosing in PACU and at the two-week follow up visit.

DETAILED DESCRIPTION:
In the last two decades, hip arthroscopy for the treatment of femoral acetabular impingement has increased rapidly. Currently, over 30k hip scopes are performed annually in the United States (incidence 1.06 per 10K). Due to anatomical differences, hip arthroscopy procedures have the potential for significant fluid extravasation when compared to knee arthroscopy. A 2011 study on hip arthroscopy showed on average 9.68 liters of fluid were used for a standard hip procedure; of that 1.13 liters absorbed into the surrounding soft tissues. A recent systematic review and meta-analysis showed warming of arthroscopic fluids significantly decreased the risk of hypothermia during hip arthroscopy. Additionally, active warming has been shown to decrease the rate of surgical site infection during numerous procedures. In total knee arthroplasty patients, a forced air warming gown significantly reduced narcotic pain consumption compared to standard care. However, the benefits of active warming for decreasing post-operative pain has not been studied in hip arthroscopy patients. Specifically, the investigators were interested in the roll the pre-warming arthroscopic fluid plays in post-operative pain after hip arthroscopy. The purpose of this study is to see if pre-warming of arthroscopic fluid reduces immediate post-surgical pain and narcotic consumption in hip arthroscopy patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18-65 years with a confirmed diagnosis of Femoroacetabular impingement (FAI)
* Required hip arthroscopy will be considered for the study
* Pre-operative history and physical exam
* Magnetic resonance imaging (MRI) before being indicated for arthroscopic surgery

Exclusion Criteria:

* Taking narcotic medications at baseline
* Have a history of complex regional pain syndrome,
* Have hip arthritis,
* Have undergone previous hip arthroscopic surgery, or
* Are deemed incapable by the Principal Investigator of completing the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Changes in Visual Analog Score | Pre-operatively, 30 and 60 minutes after completion of surgery, Post Op Days 1 and 14.
  A Visual Analog Score (VAS) will be measured pre-operatively, 30 and 60 minutes after patient arrival in the post-anesthesia care unit (PACU). Additionally, VAS will be collected in the clinic on post-operative day (POD) 1 and POD 14. The visual analog scale measures subject reported pain on a scale of 0-100 with a score of 0 indicating no pain and 100 indicating the worst pain possible.

SECONDARY OUTCOMES:
Changes in Temperature | 30-60 minutes after after completion of surgery
  Subject core temperature will be collected 30 and 60 minutes after arrival in PACU. The method for collection will be done via current standard of care.
Morphine Equivalent Dosage (MED) | After completion of surgery and at the 2-week Post Operative Visit
  Morphine equivalent dose (MED) will be calculated in PACU and at the subject's routine two-week post-operative appointment via medication reconciliation.

OTHER OUTCOMES:
Hip Outcomes Score (HOS) | Pre-operatively
  The HOS has been validated in patients with femoral acetabular impingement and has two subscales (Activities of Daily Living and Sports). The ADL subscale contained 19 items pertaining to basic daily activities, and the sports subscale contained 9 items pertaining to higher-level activities. The ADL and sports subscales are scored separately. The response to each item on the ADL subscale is scored from 4 to 0, with 4 indicating "no difficulty" and 0 indicating "unable to do." The scores for each of the items are added together to obtain a total. The total number of items with a response is multiplied by 4 to obtain the highest potential score. The item score total is divided by the highest potential score. This value is then multiplied by 100 to obtain a percentage. The sports subscale is scored in a similar manner, with the highest potential score being 36. A higher score represents a higher level of physical function.
Veterans Rand 12 (VR-12) | Pre-Operatively
  The Veterans RAND 12 Item Health Survey (VR-12) is a brief, generic, multi-use, self-administered health survey comprised of 12 items. The instrument is primarily used to measure health related quality of life and to estimate disease. The 12 items in the questionnaire correspond to eight principal physical and mental health domains including general health perceptions; physical functioning; role limitations due to physical and emotional problems; bodily pain; energy-fatigue, social functioning and mental health. The 12 items are summarized into two scores, a Physical Component Score (PCS) and a Mental Component Score (MCS). PCS and MCS summary scores are standardized using a t-score transformation and normed to a U.S. population of a score of 50 and a standard deviation of 10. The subscales are not combined or averaged for a total score. A Higher score represents a higher function.

CONTACTS AND LOCATIONS:
Overall Officials: James Genuario, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Steadman Hawkins Clinic, University of Colorado Denver, Englewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Truntzer JN, Shapiro LM, Hoppe DJ, Abrams GD, Safran MR. Hip arthroscopy in the United States: an update following coding changes in 2011. J Hip Preserv Surg. 2017 Mar 23;4(3):250-257. doi: 10.1093/jhps/hnx004. eCollection 2017 Aug. PMID 28948037
- [Background] Stafford GH, Malviya A, Villar RN. Fluid extravasation during hip arthroscopy. Hip Int. 2011 Nov-Dec;21(6):740-3. doi: 10.5301/HIP.2011.8845. PMID 22117260
- [Background] Steelman VM, Chae S, Duff J, Anderson MJ, Zaidi A. Warming of Irrigation Fluids for Prevention of Perioperative Hypothermia During Arthroscopy: A Systematic Review and Meta-analysis. Arthroscopy. 2018 Mar;34(3):930-942.e2. doi: 10.1016/j.arthro.2017.09.024. Epub 2017 Dec 6. PMID 29217304
- [Background] Ousey K, Edward KL, Lui S, Stephenson J, Walker K, Duff J, Leaper D. Perioperative, local and systemic warming in surgical site infection: a systematic review and meta-analysis. J Wound Care. 2017 Nov 2;26(11):614-624. doi: 10.12968/jowc.2017.26.11.614. PMID 29131754
- [Background] Benson EE, McMillan DE, Ong B. The effects of active warming on patient temperature and pain after total knee arthroplasty. Am J Nurs. 2012 May;112(5):26-33; quiz 34, 42. doi: 10.1097/01.NAJ.0000414315.41460.bf. PMID 22546733

DOCUMENTS (1):
  • Informed Consent Form (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/66/NCT03453866/ICF_000.pdf